CLINICAL TRIAL: NCT01513421
Title: Active Versus Non Active Drainage for the Treatment of Infected Intra-abdominal Collection: a Randomized Prospective Trial
Brief Title: Active Versus Non Active Drainage for the Treatment of Infected Intra-abdominal Collection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dr. Emmanuel Melloul, Surgeon, M.D., Centre Hospitalier Universitaire Vaudois
Other Study IDs: 281/10
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Surgery; Pancreatitis; Diverticulitis; Appendicitis
Keywords: Infected; Intra-abdominal; Collection; Drainage; Percutaneous
MeSH Terms: conditions — Pancreatitis; Diverticulitis; Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Active vacuum pressure drainage
  Interventions: Procedure: Percutaneous drainage of intra-abdominal collection
- Free drainage
  Interventions: Procedure: Percutaneous drainage of intra-abdominal collection

INTERVENTIONS:
Procedure: Percutaneous drainage of intra-abdominal collection — Percutaneous drainage of infected intra-abdominal collection Under computed tomography or ultrasound guidance.
  Procedures perform by a board certified interventional radiologist
  Other Names: Intra-abdominal drainage; Postoperative collection

SUMMARY:
The Percutaneous drainage of symptomatic intra-abdominal collection (primary or secondary to surgery)is the treatment of choice in the absence of peritonitis signs. In critically ill patients, this procedure allows to avoid or postpone surgery. In these settings, the percutaneous drain can be either in Active Vacuum Pressure or in Free drainage. However, no prospective trials has assessed the efficiency of these two modalities of drainage in cases of infected intra-abdominal collections. The investigators aimed then to prospectively analyzed the efficiency (in term of infectious control) of drainage under active vacuum pressure vs. free drainage for the treatment of infected intra-abdominal collections.

ELIGIBILITY:
Inclusion Criteria:

* Infected intra-abdominal collection requiring a percutaneous drainage after surgery or due to a primary intra-abdominal infectious disease (e.g. diverticulitis, appendicitis)
* age over 18 years old
* intra-abdominal collections >5 cm in diameter with signs of infections on imaging

Exclusion Criteria:

* pregnancy
* age< 18 years
* signs of peritonitis
* Intensive care unit patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-hospital patients with infected intra-abdominal collection (primary or secondary to surgery)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
time of drainage | 90 days after drianage

SECONDARY OUTCOMES:
Control of infection | up to 7 days after drainage
Timing of antibiotherapy | up to 15 days after drainage
Hospital stay | up to 90 days after drainage
Morbidity related to the procedure | up to 90 days after drainage
in-hospital mortality | up to 90 days after the drainage

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Melloul, M.D., Principal Investigator — Department of Visceral surgery (CHUV); Nicolas Demartines, M.D., Study Chair — Department of Visceral surgery (CHUV); Alban Denys, M.D., Study Chair — Department of Interventional radiology (CHUV)
Locations (1):
- Department of Visceral surgery, CHUV, Lausanne, Canton of Vaud, Switzerland